CLINICAL TRIAL: NCT00739050
Title: Effect of Simvastatin on Endothelial Function in Premenopausal Women With Systemic Lupus Erythematosus
Brief Title: Effect of Simvastatin on Endothelial Function in Premenopausal Women With Systemic Lupus Erythematosus (0733-271)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0733-271; 2008_021
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2010-12-16 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Arm 1: Drug
  Interventions: Drug: simvastatin
- 2 (Placebo Comparator): Arm 2: Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: simvastatin — simvastatin 20mg daily at nights for 12 weeks. Tablets
  Other Names: Zocor; MK0733
  Arms: 1
Drug: Comparator: Placebo — placebo daily at nights for 12 weeks. Tablets
  Arms: 2

SUMMARY:
Women with Systemic Lupus Erythematosus (SLE) are prone to cardiovascular disease. Early detection of improvement of endothelial function with simvastatin could be a clue for future intervention trials.

ELIGIBILITY:
Inclusion Criteria:

* Female Patients Over 18 Years Old
* Confirmed Systemic Lupus Erythematosus (SLE) diagnosis according to American College of Rheumatology (ACR)
* Signed Informed Consent Form (ICF)

Exclusion Criteria:

* Patients With LDL-C Below 90 mg/dL
* Pregnant Or Breast Feeding
* Diabetes Mellitus
* Or Any Clinically Relevant Organ Disfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-09-19 (Actual); Primary Completion 2008-02-01 (Actual); Study Completion 2008-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled (FPE): 19 Sept 2007; Last patient enrolled (LPE) 22 Oct 2007. The protocol was terminated for Administrative Reasons
Groups:
- Simvastatin: simvastatin 20 mg daily at nights for 12 weeks
- Placebo: Placebo daily at nights for 12 weeks
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 4 | 0
Completed | 3 (These 3 patients completing treatment did not complete the required procedures during the trial.) | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All Randomized patients.
  Laboratory values were only avaliable for 3 participants for Total Cholesterol, Low Density Lipoprotein Cholesterol (LDL-C), and High Density Lipoprotein Cholesterol (HDL-C)
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — N=3 (Completed Participants)
  mg/dL | 176.67 (28.50)
Low Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — N=3 (Completed Participants)
  mg/dL | 105 (23.64)
High Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — N=3 (Completed Participants)
  mg/dL | 53 (10.15)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Endothelial Thickness After 12 Weeks of Treatment.
Description: The study was terminated; no outcome measure data analyses were conducted.
Time Frame: Baseline and 12 weeks
Population: The study was terminated; no outcome measure data analyses were conducted. The Investigator was not able to recruit the required patients and was not able to get the necessary Computed Tomography equipment.
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Total Cholesterol From Baseline at Week 12
Description: The study was terminated; no outcome measure data analyses were conducted.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) After 12 Weeks of Treatment
Description: The study was terminated; no outcome measure data analyses were conducted.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) After 12 Weeks of Treatment
Description: The study was terminated; no outcome measure data analyses were conducted.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

LIMITATIONS AND CAVEATS:
The Investigator was not able to recruit the required patients and was not able to get the necessary equipment. The protocol was terminated for Administrative Reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.